CLINICAL TRIAL: NCT07364435
Title: The Effect of Two Different Bed Bathing Methods on Vancomycin-Resistant Enterococcus Colonization in Intensive Care Patients: A Randomized Controlled Trial
Brief Title: Effect of Bed Bathing Methods on VRE Colonization in ICU Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Özkan Kasap (Other Government)
Responsible Party: Sponsor-Investigator, Özkan Kasap, Nurse, Başakşehir Çam & Sakura City Hospital
Organization: Başakşehir Çam & Sakura City Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024-188
Record Dates: First submitted 2026-01-16; First posted 2026-01-23 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Vancomycin-Resistant Enterococcus
MeSH Terms: interventions — Chromogranins; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4% Chlorhexidine Gluconate Bed Bath (Experimental): Participants receive daily whole-body bed bathing using a 4% chlorhexidine gluconate solution as part of the bed bathing procedure.
  Interventions: Procedure: Bed Bath; Drug: Chlorhexidine gluconate 4%
- Disposable Antibacterial Bed Bath Wipes (Active Comparator): Participants receive daily bed bathing using disposable antibacterial body cleansing wipes.
  Interventions: Device: Disposable antibacterial bed bath wipes

INTERVENTIONS:
Procedure: Bed Bath — Daily whole-body bed bathing performed as part of routine ICU care.
  Other Names: Daily whole-body bathing with 4% chlorhexidine gluconate solution.
  Arms: 4% Chlorhexidine Gluconate Bed Bath
Device: Disposable antibacterial bed bath wipes — Daily whole-body bed bathing using disposable antibacterial body cleansing wipes as part of routine ICU care.
  Other Names: Daily bed bathing using disposable antibacterial body cleansing wipes.; Antibacterial bathing wipes
  Arms: Disposable Antibacterial Bed Bath Wipes
Drug: Chlorhexidine gluconate 4% — A 4% chlorhexidine gluconate solution used during the bed bathing procedure for whole-body skin antisepsis in ICU patients.
  Other Names: CHG 4% solution
  Arms: 4% Chlorhexidine Gluconate Bed Bath

SUMMARY:
This randomized controlled trial aims to compare the effects of two different bed bathing methods on vancomycin-resistant Enterococcus (VRE) colonization in adult intensive care unit patients. A total of 210 patients were randomly assigned to receive either daily whole-body bathing with 4% chlorhexidine gluconate solution or daily bed bathing using disposable antibacterial body wipes. VRE colonization was monitored using skin swab cultures collected on days 7, 14, and 21. The results of this study may contribute to infection prevention strategies in intensive care units by identifying effective hygiene practices for reducing VRE colonization.

DETAILED DESCRIPTION:
This study was designed as a randomized controlled trial conducted in the general intensive care units of a tertiary care hospital. Adult patients meeting the inclusion criteria were randomly assigned to one of two parallel groups. The experimental group received daily whole-body bed bathing with a 4% chlorhexidine gluconate solution, while the control group received daily bed bathing using disposable antibacterial body cleansing wipes.

Randomization was performed to ensure comparable baseline characteristics between the groups. VRE colonization was assessed through skin swab cultures obtained at baseline and subsequently on days 7, 14, and 21. The primary outcome of the study was the rate of VRE colonization over time. Secondary analyses included the evaluation of patient-related factors such as age, length of stay, body mass index, and previous VRE history.

All procedures were performed by trained nursing staff according to standardized protocols. The study was conducted following ethical approval obtained from the institutional ethics committee, and informed consent was obtained in accordance with ethical standards. The findings of this study aim to support evidence-based infection control practices in intensive care nursing.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years and older
* Patients admitted to the intensive care unit
* Expected ICU stay of at least 48 hours
* Patients requiring daily bed bathing

Exclusion Criteria:

* Known hypersensitivity to chlorhexidine
* Extensive skin lesions or burns
* Patients colonized or infected with VRE at ICU admission
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Vancomycin-Resistant Enterococcus (VRE) Colonization | Baseline, Day 7, Day 14, and Day 21
  The presence of vancomycin-resistant Enterococcus (VRE) colonization assessed by skin swab cultures obtained from intensive care unit patients. Cultures were collected at baseline and on days 7, 14, and 21 to compare the effect of two different bed bathing methods.

SECONDARY OUTCOMES:
Change in VRE Colonization Over Time | Day 7, Day 14, and Day 21
  Changes in VRE colonization status over time were evaluated to assess the temporal effect of bed bathing methods during intensive care unit stay.

CONTACTS AND LOCATIONS:
Overall Officials: Ayfer Ozbas, Prof.Dr., Principal Investigator — T.C. DEMIROGLU SCIENCE UNIVERSITY
Locations (1):
- Basaksehir Pine and Sakura City Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. This study was conducted as a single-center academic randomized controlled trial, and the informed consent and ethics committee approval did not include provisions for public data sharing. All data are analyzed and reported in aggregate form to protect participant confidentiality.